CLINICAL TRIAL: NCT05272553
Title: Investigating the Application of Narrative Exposure Therapy (NET) to Reduce Symptoms of Traumatic Stress in Cancer Patients Not in Active Treatment: a Naturalistic Single Case Study Series
Brief Title: Narrative Exposure Therapy to Reduce Symptoms of Traumatic Stress in Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21083
Record Dates: First submitted 2022-01-06; First posted 2022-03-09 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Stress Disorder; Cancer
Keywords: narrative exposure therapy
MeSH Terms: conditions — Stress Disorders, Traumatic; Neoplasms

STUDY DESIGN:
Intervention Model Description: Naturalistic, mixed-method, explanatory sequential measurement single case series design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative Exposure Therapy (Experimental): This is a single case series design which focuses on assessing whether Narrative Exposure Therapy could reduce symptoms of traumatic stress in cancer survivors; no comparator will be included.
  Interventions: Other: Narrative Exposure Therapy

INTERVENTIONS:
Other: Narrative Exposure Therapy — NET (Schauer et al., 2011) is an evidence-based, short-term, manualised treatment for trauma-spectrum disorders; it aims to reduce symptoms of traumatic stress in individuals who continue to suffer from past experiences of traumatic stressors; NET combines principles of CBT, Testimony Therapy, and Exposure Therapy.

SUMMARY:
The main purpose of the study is to evaluate the feasibility, acceptability, and potential effectiveness of NET in reducing symptoms of traumatic stress (e.g., hyperarousal, avoidance, and intrusion) in cancer patients who are not in active treatment.

Further aims include:

* Can NET be effective in reducing symptoms of existential anxiety, anxiety, and depression in cancer patients who are not in active treatment?
* Can NET improve the Quality of Life (QoL) of cancer patients who are not in active treatment? And are improvements in QoL associated to reduction of traumatic stress?
* Can NET lead to post-traumatic growth?
* Does the NET protocol need to be adapted to meet cancer patients' needs?

DETAILED DESCRIPTION:
Research has shown that cancer can lead to significant emotional and social distress. Many elements of the cancer experience can be perceived as traumatic by cancer patients, including diagnostic testing, waiting periods, prolonged and invasive treatment procedures, follow-up scans, and fear of recurrence.

Unlike single traumatic events, cancer behaves as an ongoing and chronic stressor. Emotional and social distress (including anxiety, depression, and post-traumatic stress disorders), can lead to reduced treatment compliance and less adherence to a healthy lifestyle which might compromise chances of survival.

Research has shown that due to the psychological distress experienced during diagnosis, treatment, and survivorship, cancer patients are interested in receiving psychosocial support; unfortunately, their distress is often perceived as "normal" and "manageable" by professionals. The result is that 30-40% of cancer patients are not supported.

This study aims to evaluate whether Narrative Exposure Therapy (NET) can be a feasible, acceptable, and effective intervention to reduce symptoms of traumatic stress in adult cancer patients who are not in active treatment. NET is a time-limited, structured, and evidenced-based intervention designed to reduce symptoms of traumatic stress through two main processes: fear habituation and integration of the traumas within the autobiographical memory. Six participants will be recruited with the support of Clinical Psychologists working in cancer services across Nottinghamshire and Lincolnshire, they will receive around twelve weekly interventions sessions. Changes will be explored through outcome measures administered before, during, and after the intervention and through interviews about their experience at the end.

The study is founded by The University of Nottingham. Potential benefits include providing initial evidence to address traumatic stress in cancer patients, providing an intervention which could be suitable for psycho-oncology services which might lack resources to offer long-term psychosocial support, and contributing to the evidence for the use of NET in a new group.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 and over)
* Diagnosed with cancer in adulthood
* Able to provide informed consent
* Able to communicate verbally and speak English
* Not in active treatment (at any stage post-treatment)
* Suffer from symptoms of traumatic stress caused or triggered by the cancer experience. A diagnosis of PTSD is not required (PTSD Checklist Civilian, PCL-C cut-off score: 29 and above).
* No specific form of cancer

Exclusion Criteria:

Participants have a known diagnosis of Intellectual Disability (ID)

* Participants must not be receiving other forms of psychosocial support whilst engaging in NET
* They are substance dependent
* They are actively psychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in PTS symptoms between the baseline, NET intervention, and 1 month and up to three months follow-up phases - as assessed by thePTSD Checklist - Civilian (PCL-C; Weathers et al., 1994) | Throughout the study, for approximately 31 weeks
  The PCL-C explores items related to individuals' past stressful experiences using a 17-item self-report checklist (Weathers et al., 1994). The PCL-C has been widely used in cancer research (such as DuHamel et al., 2010; Levine et al., 2005; Lleras de Frutos et al., 2020; Ochoa-Arnedo et al., 2020) and was assessed as a screening instrument by Andrykowski and colleagues in their study with breast cancer survivors in 1998. The PCL-C has shown good internal consistency (Cronbach's alpha >.75) (Wilkins et al., 2011) and good test-retest reliability with scores ranging from 0.68 and 0.92 (Hahn et al., 2015). Scores above 29 are indicative of clinical concerns; the US Department of Veterans Affairs recommends a cut-off score of 30 to 38 for diagnosis of PTSD (www.ptsd.va.gov).

SECONDARY OUTCOMES:
Change in depression and anxiety symptoms between the baseline, NET intervention, and 1 month and up to three months follow-up phases - as assessed byHospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983) | Throughout the study, for approximately 31 weeks
  The HADS is the most extensively studied mood scale in cancer services (as well as in other medical settings) (Mitchell et al., 2010). It is a fourteen item self-report measure of anxiety and depression that has demonstrated to be psychometrically robust showing good internal consistency (Anxiety Cronbach's alpha = .83; Depression Cronbach's alpha = .82) (Bjelland et al., 2002) and good test-retest reliability (Anxiety r = .82; Depression r = .52) (Martin & Thompson, 2002). Scores of 8 and above are indicative of clinical concerns.
Change in cancer-specific quality of life between the baseline, NET intervention, and 1 month and up to three months follow-up phases - as assessed by the Functional Assessment of Cancer Therapy - General 7 items (FACT-G7; Yanez et al., 2013) | Throughout the study, for approximately 31 weeks
  The FACT-G7 is a brief, cancer-specific quality-of-life measure comprising 7 items from the 27-item Functional Assessment of Cancer Therapy-General Scale (FACT-G; Cella et al., 1993) that were endorsed by cancer patients as being of highest priority. Its items comprise physical, emotional and functional domains. Total scores range between 0 and 28, and higher scores indicate better quality of life. The FACT-G7 has shown good internal consistency (Cronbach's alpha = between .72 and .80) (Mah et al., 2020) and good test-retest reliability (scores between .52 and .74) (King et al., 2020).

OTHER OUTCOMES:
Process measure of habituation: Subjective Unit of Distress (SUD; Wolpe, 1969) | For approximately ten weeks
  The SUD is a self-report scale from 0 to 10 for measuring the subjective intensity of distress experienced by an individual; subjective distress refers to uncomfortable or painful emotions felt. The SUD will be completed pre and post narration of each trauma event to assess for within session habituation and then repeated for re-narration of each trauma event for between session habituation.
Change in post traumatic growth between the baseline, the last NET session, and 1 month and up to three months follow up phases - as assessed by the Post-traumatic growth inventory (PTGI; Tedeschi & Calhoun, 1996) | On week two, week 15, week 19, and week 31
  Post traumatic growth is defined as the ability of the individual to experience positive changes in the aftermath of extremely negative experiences; the positive changes usually occur in the context of the self, interpersonal relationships, and philosophy of life (Anderson & Lopez-Baez, 2017). The PTGI consists of 21 items which cover five domains: relating to others, new possibilities, personal strength, spiritual change, and appreciation of life. The PTGI has shown good internal consistency (Cronbach's alpha = .90) and test-retest reliability (r = .71) (Tedeschi & Calhoun, 1996).
Change in existential anxiety symptoms between the baseline, the last NET session, and 1 month and up to three months follow up phases - as assessed by theExistential Concerns Questionnaire (ECQ; van Bruggen, 2018) | On week two, week 15, week 19, and week 31
  Existential anxiety represents a form of anxiety that goes beyond experiencing anxiety as a consequence of a concrete threat, it is instead related to a threat to our existence as a whole (Glas, 2003); as mentioned in the background section, cancer patients often question their own individual values and the meaning of their existence. Research has demonstrated that cancer patients with higher levels of existential well-being (e.g., less fear related to disease recurrence) report better QoL and lower emotional distress (Brady et al., 1999; Edmondson et al., 2008, Visser et al., 2010). This 13-item questionnaire covers anxiety in reaction to death, guilt, and meaninglessness. The ECQ has shown good internal consistency with a Cronbach's alpha of .91 and test-retest reliability (van Bruggen, 2018).
Change in body awareness and autonomic reactivity between the baseline, the last NET session, and 1 month and up to 3 months follow-up phases - as assessed by the Body Perception Questionnaire Short Form - Autonomic Nervous System (Porges, 1993, 2015) | On week two, week 15, week 19, and week 31
  The Body Perception Questionnaire (BPQ) is a self-report measure of body awareness and autonomic reactivity. For the purpose of this research project, the Autonomic Nervous System subscale was taken into consideration. The autonomic nervous system (ANS) is a set of neural pathways connecting the brain and body; these pathways send information and signals from the body about the status of organs and tissues (i.e., afferent projections). These signals can alter the functions of the body, depending on internal and external needs. The BPQ-SF has shown good internal consistency (categorical omega between .77 and .96) and test-retest reliability (r = .96 to .99).
Change Interviews (Elliot et al., 2001) | At 1 month follow up
  The feasibility and acceptability of video NET will be investigated by conducting Change Interviews with participants approximately one month after completing the treatment. In this instance, the participant will be asked to provide feedback on their experience of receiving treatment, including in terms of barriers and fascinators to engagement. The interviews will be conducted by an external researcher, i.e. another Trainee Clinical Psychologist, following an adaptation of Elliott, Slatick, & Urman's (2001) protocol. The interviews will be audio- or video-recorded and then sent to the student/investigator for transcription and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schröder, Principal Investigator — The University of Nottingham
Locations (1):
- The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No